CLINICAL TRIAL: NCT06051292
Title: Decremental Esophageal Catheter Filling Volume Titration For Esophageal Pressure Measurement
Brief Title: Decremental Esophageal Catheter Filling Volume Titration For Transpulmonary Pressure Measurement
Acronym: DECFVTTPM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Hasan ağın, Professor, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02020395
Record Dates: First submitted 2023-09-14; First posted 2023-09-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Acute Respiratory Distress Syndrome (PARDS); Acute Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: Acute respiratory failure (ARF); esophageal catheter; transpulmonary pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast decremental (Experimental): fast decremental catheter volume titration will be applied
  Interventions: Other: Fast method
- Conventional (Active Comparator): conventional catheter volume titration will be applied
  Interventions: Other: Conventional method

INTERVENTIONS:
Other: Fast method — Fast decremental catheter volume titration will be applied and optimal filling volume will be determined according to the measurements
  Arms: Fast decremental
Other: Conventional method — Conventional catheter volume titration will be applied and optimal filling volume will be determined according to the measurements
  Arms: Conventional

SUMMARY:
Mechanical ventilation is a critical intervention in the management of pediatric patients with respiratory distress. During this process, accurate measurement of transpulmonary pressure (PL) is essential to ensure the safety and efficacy of ventilation. PL is defined as the difference between alveolar pressure (Palv) and pleural pressure (Ppl). While the direct measurement of Ppl is possible, it poses a risk to tissue integrity. Thus, the primary surrogate for Ppl measurement today is esophageal pressure (Pes).

However, the measurement of Pes is not without challenges. This abstract outlines the pitfalls associated with Pes measurement, emphasizing the importance of employing well-defined procedures to mitigate potential errors. These errors can range from underestimation of Pes due to underfilled catheters to overestimation resulting from overfilled catheters.

To address these challenges and optimize Pes measurement, various methods have been proposed for titrating the filling volume of the esophageal catheter. In this study, investigators aim to assess a faster decremental filling method and compare it to the traditionally accepted Mojoli method in the context of pediatric patients. This research seeks to enhance the intensivists' understanding of the most efficient and accurate approach to Pes measurement during mechanical ventilation in the pediatric population, ultimately contributing to improved patient care and outcomes

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 1 months and 18 years
* Patients need mechanical ventilation support without modification of ventilation settings within the upcoming 2 hours
* Informed consent was signed by next of kin
* Requiring esophageal catheter application

Exclusion Criteria:

* Patients eligible for extubation or modification of ventilation settings within the upcoming 2 hours
* Patient included in another interventional study in the last 30 days
* Patients unable to undergo esophageal catheter insertion due to congenital or acquired pathologies
* Patient included in another interventional research study under consent
* Patient already enrolled in the present study in a previous episode of acute respiratory failure

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Optimal catheter filling volume | up 1 hour after catheter placement
  The clinician will determine the optimal filling volume of the catheter using two distinct methods

SECONDARY OUTCOMES:
Transpulmonary driving pressure | up 1 hour after catheter placement
  The measured transpulmonary driving pressure achieved using the optimal filling volume of the catheter
Time | up 1 hour after catheter placement
  The duration necessary to ascertain the optimal filling volume of the esophageal catheter

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Agin, Professor, Study Director — Behcet Uz Children's Hospital
Locations (4):
- Turkey (Türkiye) (4):
  - Aydin Obstetric and pediatrics Hospital, Aydin
  - Erzurum Regional Research and Training Hospital, Erzurum
  - Cam Sakura Research and Training Hospital, Istanbul
  - The Health Sciences University Izmir Behçet Uz Child Health and Diseases Research and Training Hospital, Izmir

REFERENCES:
- [Background] Mojoli F, Chiumello D, Pozzi M, Algieri I, Bianzina S, Luoni S, Volta CA, Braschi A, Brochard L. Esophageal pressure measurements under different conditions of intrathoracic pressure. An in vitro study of second generation balloon catheters. Minerva Anestesiol. 2015 Aug;81(8):855-64. Epub 2015 Jan 30. PMID 25634481
- [Background] Hotz JC, Sodetani CT, Van Steenbergen J, Khemani RG, Deakers TW, Newth CJ. Measurements Obtained From Esophageal Balloon Catheters Are Affected by the Esophageal Balloon Filling Volume in Children With ARDS. Respir Care. 2018 Feb;63(2):177-186. doi: 10.4187/respcare.05685. Epub 2017 Oct 31. PMID 29089460
- [Background] Mojoli F, Iotti GA, Torriglia F, Pozzi M, Volta CA, Bianzina S, Braschi A, Brochard L. In vivo calibration of esophageal pressure in the mechanically ventilated patient makes measurements reliable. Crit Care. 2016 Apr 11;20:98. doi: 10.1186/s13054-016-1278-5. PMID 27063290